CLINICAL TRIAL: NCT07313111
Title: Efficacy of Thymoquinone as an Adjuvant Treatment With Pregabalin for the Treatment of Neuropathy in Diabetic Patients: A Randomized Clinical Trial of 65 mg of Thymoquinone and 75 mg Pregabalin Daily for Two Months
Brief Title: Thymoquinone as an add-on Therapy for the Management of Patients With Diabetic Peripheral Neuropathy
Acronym: TQDPN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Nermin Jamal Abdulqadr, assistant lecturer Msc Pharmacology, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HawlerMU-1; HawlerMU-TQPG_2025 (Other: Hawler Medical University, College of Medicine)
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)
Keywords: diabetic neuropathy; thymoquinone; nerve conductive study; oxidative stress
MeSH Terms: conditions — Diabetic Neuropathies | interventions — thymoquinone

STUDY DESIGN:
Intervention Model Description: Group one received standard treatment (pregabalin) and group two received standard treatment plus interventional treatment (pregabalin + thymoquinone)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (stander treatment only Pregabalin) (Active Comparator): Participants in this arm received 75 mg of pregabalin capsule orally for two months
  Interventions: Drug: stander treatment pregabalin
- supplement (thymoquinone)+ standard treatment (pregabalin) (Experimental): participants in this arm received thymoquinone capsule 65 mg + pregabalin capsule 65 mg daily for two months
  Interventions: Drug: stander treatment pregabalin; Dietary Supplement: thymoquinone

INTERVENTIONS:
Drug: stander treatment pregabalin — Participants received 75 mg of a pregabalin capsule for two months
Dietary Supplement: thymoquinone — participants recieved 65 mg of thymoquinone capsule daily for two months
  Arms: supplement (thymoquinone)+ standard treatment (pregabalin)

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of thymoquinone as an adjuvant treatment with pregabalin in the management of diabetic peripheral neuropathy for both sexes older than 18 years.

The main questions it aims to answer are:

* Whether the use of thymoquinone could improve diabetic neuropathy and be confirmed by a nerve conduction study?
* Could thymoquinone improve oxidative stress and inflammation by using these parameters (visfatin, calprotectin, malondialdehyde)?
* Does thymoquinone improve neuropathic pain by using the VAS scale for pain?

DETAILED DESCRIPTION:
Study Design and Methodology This is a randomized, clinical trial designed to evaluate the neuroprotective effects of thymoquinone in diabetic patients with neuropathy.

Study Sites Primary Location: Galyawa diabetic center and Neurophysiology Department of Hawler Psychiatric Hospital, affiliated with Hawler Medical University.

Multicenter expansion was considered, but all participants were recruited at the primary site.

Study Population Enrollment (Actual): 50 participants with diabetic neuropathy Groups: Group 1 (n=25): DPN patients on Pregabalin 75 mg daily for 2 months. Group 2 (n=25): DPN patients on Pregabalin 75 mg + Thymoquinone 65 mg daily for 2 months.

Follow-up Period Duration: 2 months from initiation of treatment. Assessment intervals: Baseline (pre-treatment) and 2 months (post-treatment). Primary outcome: A Nerve conductive study was done, and blood samples for (visfatin, calprotectin, malondialdehyde, and HbA1c) measurement were drawn before starting treatment.

Secondary or Endpoints: the same investigations were done after two months of treatment Adverse Events: Monitored continuously throughout the 2-month treatment and follow-up, including risks of epigastric pain, dizziness, and headache.

Statistical Analysis Plan Sample Size: Originally planned for 80 patients, but 50 were enrolled (25 per group).

Comparative Analysis: Paired t-tests, Wilcoxon signed-rank tests (for non-parametric data), ANOVA for repeated measures where appropriate.

Ethical Considerations Approved by the Hawler Medical University Ethics Committee.

Written informed consent was obtained from all participants. Potential Impact: If thymoquinone proves effective, this study could support the use of thymoquinone as a neuroprotective strategy in diabetic neuropathic patients, improving NCS outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Both males or females of any race over 18 years of age.
2. Patients with either type1 or type2 diabetes, who have been on a stable anti-diabetic medication regimen for at least 30 days before randomization.
3. Duration of painful diabetic peripheral neuropathy was required to be more than 3 months.

Exclusion Criteria:

1. History of smoking, alcohol consumption, and thyroid gland disorder.
2. Patients with any kidney disorder or any conditions that could confound the assessment of pain due to diabetic peripheral neuropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
peripheral nerve improvement through NCS | Evaluated at base time (before treatment) and two months after treatment
  NCS assessment of both upper and lower limbs to detect diabetic neuropathy, including measurement tools: latency, amplitude, and conduction velocity for motor and sensory nerves.

SECONDARY OUTCOMES:
oxidative stress, and inflammatory parameter levels | Evaluated at baseline (before treatment) and two months after treatment
  Measurement of serum Visfatin, Calprotectin, Malondialdehyde, and HbA1c for all participants

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler medical university, Galyawa diabetic center and Neurophysiology department of hawler psychiatric hospital, Erbil, IRAQ, Iraq

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared publicly. The data will be kept confidential to ensure participant privacy and comply with ethical and regulatory requirements, including those related to informed consent and data protection. Access to the data may be considered for future collaborations under strict ethical guidelines and approval from the relevant oversight bodies.